CLINICAL TRIAL: NCT01252797
Title: RAD 1002: Phase I Dose Escalation/De-escalation Study of Pre-operative Stereotactic Radiosurgery for Brain Metastases
Brief Title: Dose Escalation/De-escalation Study of Pre-operative Stereotactic Radiosurgery for Brain Metastases(RAD 1002)
Acronym: RAD 1002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Fiveash, MD, Professor and Vice Chair, University of Alabama at Birmingham Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F100528006
Record Dates: First submitted 2010-11-22; First posted 2010-12-03 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Brain Metastases
Keywords: brain metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stereotactic Radiosurgery (15 Gy) (Active Comparator): Group A: If the tumor which will be surgically removed is at least 2 cm and up to 4 cm in maximum diameter, then this group will receive Dose Level II (15 Gy) of radiation: stereotactic radiosurgery (SRS) followed by surgery to remove the tumor.
  Interventions: Radiation: Stereotactic Radiosurgery (15 Gy)
- Stereotactic Radiosurgery (12Gy) (Experimental): Group B: If the tumor which will be surgically removed is larger than 4 cm and up to 6 cm in diameter, then this group will receive Dose Level I (12 Gy) of radiation: stereotactic radiosurgery (SRS) followed by surgery to remove the tumor.
  Interventions: Radiation: Stereotactic Radiosurgery (12 Gy)

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (15 Gy) — Group A will start at dose level II: 15 Gy
  Group B will start at dose level I: 12 Gy
  Arms: Stereotactic Radiosurgery (15 Gy)
Radiation: Stereotactic Radiosurgery (12 Gy) — Group B will start at Dose Level I: 12 Gy
  Arms: Stereotactic Radiosurgery (12Gy)

SUMMARY:
This study will investigate the safety, tolerability, and effectiveness of changing the order of receiving radiation therapy for treating brain cancer. The investigators hope that changing the sequence of radiation therapy will lower the risk of cancer spreading throughout your spinal fluid, which covers your brain and spinal cord.

DETAILED DESCRIPTION:
This study will attempt to determine the maximum tolerated dose of pre-operative stereotactic radiosurgery (SRS) in the treatment of brain metastases. Patients will be placed in one of two dose groups based on index tumor size, and dose will be adjusted according to presence or absence of dose limiting toxicity (DLT).

Group A: Index Tumor > 2 cm and up to 4 cm in maximum diameter Group B: Index Tumor > 4 cm and up to 6 cm in maximum diameter

Dose escalation or de-escalation will be conducted via a modified 3+3 method at the following levels. Group A will start at dose level II. Group B will start at dose level I.

Dose Level I: 12 Gy Dose Level II: 15 Gy

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have history of histologically confirmed malignancy. Brain biopsy is not required unless diagnosis is judged to be in doubt by the treating physician.
* Newly diagnosed brain metastases (four or fewer by post-contrast MRI obtained within six weeks of study entry)
* At least one brain metastasis (index tumor) must be within 2-6 cm in maximum diameter and deemed appropriate for surgical resection by the treating neurosurgeon.
* Karnofsky performance status (KPS) of greater than or equal to 60
* Age greater than 19
* Life expectancy greater than 12 weeks
* Subjects given written informed consent

Exclusion Criteria:

* Patients with small cell lung cancer and lymphoma are ineligible.
* More than four metastases by baseline post-contrast MRI
* Prior whole brain radiation therapy
* Insufficient recovery from all active toxicities of prior therapies
* Subjects who are deemed to be poor surgical risks by the treating neurosurgeon because of medical comorbidities
* Pregnant or nursing women
* Women of childbearing potential who are not using an effective method of contraception are excluded. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to administration of SRS.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2016-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of preoperative stereotactic radiosurgery (SRS) for brain metastasis | one year
  The maximum tolerated dose (MTD) is defined as the highest dose of stereotactic radiosurgery delivered pre-operative at which no more than 2 out of 6 patients experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Acute Toxicity with preoperative stereotactic radiosurgery (SRS) | 6 months
  Any possible, probable, or definite treatment-related AE or SAE (assessed by CTCAE 4.0) occurring within six months or less from the date of stereotactic radiosurgery was received.
Late Toxicity with preoperative stereotactic radiosurgery (SRS) | 1 year
  Any possible, probable, or definite treatment-related AE or SAE (assessed by CTCAE 4.0) occurring more than six months from the date of stereotactic radiosurgery was received.
Rates of Local Control | 2 years
  This will be assessed by MRI Imaging obtained post-operatively at follow-up visits.
Rates of Leptomeningeal Dissemination | 2 years
  Leptomeningeal Dissemination (LMD) defined as diffuse carcinomatosis and/or distant focal pachymeningeal (dural) tumor and assessed by MRI Imaging for the study period.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Fiveash, MD, Principal Investigator — Hazelrig-Salter Radiation Oncology Center (HSROC)/ University of Alabama at Birmingham (UAB)
Locations (1):
- Hazelrig-Salter Radiation Oncology Center/University of Alabama at Birmingham, Birmingham, Alabama, United States